CLINICAL TRIAL: NCT02734667
Title: Initiation of Continuous Glucose Monitoring at Diagnosis of Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korey Hood (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor-Investigator, Korey Hood, Clinical Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35990
Record Dates: First submitted 2016-03-09; First posted 2016-04-12 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CGM at diagnosis of T1D (Experimental): Participants start non-adjunctive use of CGM at diagnosis of T1D and continue for 6 months.
  Interventions: Device: CGM at diagnosis of T1D
- Usual Care (No Intervention): Participants receive usual care for T1D for 6 months post diagnosis.

INTERVENTIONS:
Device: CGM at diagnosis of T1D — Initiation of non-adjunctive CGM use at diagnosis of T1D
  Arms: CGM at diagnosis of T1D

SUMMARY:
The purpose of this study is to learn about the impact of continuous glucose monitoring (CGM) on families with newly diagnosed children with type 1 diabetes (T1D). The investigators hope to learn about how continuous glucose monitoring affects glycemic variables and diabetes-related distress.

DETAILED DESCRIPTION:
Synopsis of study protocol

This pilot randomized clinical trial compares newly diagnosed T1D youth who are started on CGM (the intervention group) versus those who are not (the control group). The investigators will examine group differences over a 6-month period (Phase 1) on two sets of outcomes: psychosocial variables and glycemic variables. After the initial comparison of intervention to control across the first six months after diagnosis, the investigators will conduct a longitudinal follow-up (Phase 2) of glycemic and psychosocial variables for an additional 18 months. The CGM system used in this study is the Dexcom G5 System with the Share function (FDA Approved). An IDE was obtained to use this system in a non-adjunctive manner. Participants will complete Phase 1 in six months. Phase 2 includes 3 more assessments conducted every six months until participants are two years post-diagnosis.

Study Procedures

Participants will be recruited at two centers: Stanford University and the Barbara Davis Center for Diabetes, University of Colorado. Participants will be enrolled while inpatient or within 1 month of diagnosis. Once identified, study staff will approach potential participants to explain the study, determine eligibility, and obtain informed consent. Once enrolled in the study, participants will be randomized. Participants will be randomized at a 2:1 ratio, intervention to control. The investigators will also stratify by age group to ensure equal representation of ages across groups. The age groups (in years) are 2-6, 7-11, and 12-17. To ensure safety in the youngest group, recruitment of participants in the age 2-6 years group will not begin until the investigators have at least 2 weeks of non-adjunctive CGM use data in at least 3 participants aged 7-17 years. Data will be reviewed by the DSMB on these 3 participants and if deemed safe by the DSMB, the investigators will start enrolling participants in the youngest age group.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, a child must meet the following criteria:

1. Diagnosis of type 1 diabetes according to American Diabetes Association diagnostic criteria
2. Time since diagnosis of no longer than one month
3. Age between 2 and 17 years
4. Parental consent (and assent from the child where applicable) to participate in the study
5. No severe medical conditions, which in the opinion of the investigators are likely to hinder participation in this clinical trial.

To be eligible for the study, a parent must meet the following criteria:

1. Parent or legal guardian of a child with type 1 diabetes meeting the "child" criteria outlined above
2. Age of 18.0 years or older
3. Parent comprehends written English
4. Parent understands the study protocol and signs the informed consent document

Exclusion Criteria:

The presence of any of the following is an exclusion for the study:

1. Child has a medical disorder that in the judgment of the investigator will interfere with completion of any aspect of the protocol (e.g., pregnancy, kidney disease, adrenal insufficiency, skin condition that may hinder sensor application).
2. Child has a neurologic disorder that in the judgment of the investigator will affect completion of the protocol
3. Current use of oral glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study
4. Child is unable to completely avoid acetaminophen for duration of study

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2016-02; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Korey K Hood, PhD, Principal Investigator — Stanford University; Bruce Buckingham, MD, Principal Investigator — Stanford University; Paul Wadwa, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Both youth and parent were enrolled; parents were enrolled for assessments of surveys only, youth under 11 years of age did not complete surveys.
Groups:
- CGM at Diagnosis of T1D: Participants start non-adjunctive use of continuous glucose monitoring (CGM) at diagnosis of type 1 diabetes (T1D) and continue for 6 months.
  CGM at diagnosis of T1D: Initiation of non-adjunctive CGM use at diagnosis of T1D
  Both groups followed through for up to 24 months
- Usual Care: Participants receive usual care for T1D for 6 months post diagnosis.
  Both groups followed through for up to 24 months
Period: Overall Study
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Started | 84 | 36
Youth | 42 | 18
Parent | 42 | 18
Completed | 82 | 30
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Population: Only youth were assessed for baseline characteristics.
Groups:
- CGM at Diagnosis of T1D: Participants start non-adjunctive use of CGM at diagnosis of T1D and continue for 6 months.
  CGM at diagnosis of T1D: Initiation of non-adjunctive CGM use at diagnosis of T1D
  Both groups followed through for up to 24 months
- Total: Total of all reporting groups
Arm/Group | CGM at Diagnosis of T1D | Usual Care | Total
Number analyzed (Participants) | 42 | 18 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 18 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.23 (3.58) | 10.30 (3.51) | 10.95 (3.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 4 | 28
  Male | 18 | 14 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 38 | 16 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 18 | 60

OUTCOME MEASURES:

1. Primary Outcome: Time Spent in Blood Glucose Range (70-180mg/dL)
Description: Increasingly it is recognized that the percent time spent in a target blood glucose range, which is set by the American Diabetes Association, is an important outcome. This measure will be used as a primary outcome and derived from objective data downloads. It is calculated using the values for 14 days around the assessment time point.
Time Frame: Collected entire period for 6 months post-baseline; primary endpoint is 14 day period around that 6-month time point
Population: This outcome was assessed in youths only.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 42 | 18
percentage of time | 64.99 (18.39) | 62.54 (19.10)
Statistical Analysis 1: Comparison: CGM at Diagnosis of T1D vs Usual Care; Test type: Superiority; p = 0.64, Regression, Linear — Generalized linear models were used to compare outcomes between the CGM and control groups at 6 months while adjusting for participant gender, age, annual household income, days since diagnosis, and baseline A1c; t statistic from GLM/regression = -0.47

2. Primary Outcome: Glucose Monitoring Satisfaction Survey (GMSS) - Parent
Description: The GMSS is a validated survey created to measure the level of satisfaction a person with diabetes - type 1 or type 2 - experiences in response to monitoring glucose values. It was validated in people using CGM. Scores range 0 to 5 with higher scores indicating greater satisfaction.
Time Frame: Baseline, 24 months
Population: Participants with complete data (by youth and parent) are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 49 | 21
score on a scale
  Youth - baseline: number analyzed (Participants) | 17 | 7
  Youth - baseline | 3.52 (0.50) | 3.54 (0.27)
  Youth - 24 months: number analyzed (Participants) | 17 | 7
  Youth - 24 months | 3.76 (0.6) | 3.82 (0.54)
  Parent - baseline: number analyzed (Participants) | 32 | 14
  Parent - baseline | 3.65 (0.59) | 3.28 (0.68)
  Parent - 24 months: number analyzed (Participants) | 32 | 14
  Parent - 24 months | 3.91 (0.66) | 3.75 (0.77)
Statistical Analysis 1: Comparison: CGM at Diagnosis of T1D vs Usual Care; Test type: Superiority; p = 0.013, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; t-statistic from GLM/regression results = -2.60

3. Primary Outcome: Time Spent in Hypoglycemia (< 70 mg/dL)
Description: Time spent in hypoglycemia is calculated using the values for 14 days around the assessment time point.
Time Frame: Collected entire period for 6 months post-baseline; primary endpoint is 14 day period around that 6-month time point
Population: This outcome was assessed in youths only.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 42 | 18
percentage of time | 1.87 (1.65) | 5.06 (5.13)
Statistical Analysis 1: Comparison: CGM at Diagnosis of T1D vs Usual Care; Test type: Superiority; p = 0.003, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; t-statistic from GLM/regression results = 3.12

4. Secondary Outcome: Pediatric Quality of Life Inventory
Description: This is a measure of health-related quality of life. It is used to understand the broader impact on quality of life which includes social, psychological, and health aspects of daily living. Scores range from 0 to 100. Higher scores indicate greater quality of life.
Time Frame: Baseline, 24 months
Population: Participants with complete data (by youth and parent) are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 49 | 21
score on a scale
  Youth - baseline: number analyzed (Participants) | 17 | 7
  Youth - baseline | 75.38 (13.48) | 85.23 (8.25)
  Youth - 24 months: number analyzed (Participants) | 17 | 7
  Youth - 24 months | 82.67 (14.49) | 92.08 (10.31)
  Parent - baseline: number analyzed (Participants) | 32 | 14
  Parent - baseline | 75.27 (14.79) | 81.05 (12.26)
  Parent - 24 months: number analyzed (Participants) | 32 | 14
  Parent - 24 months | 81.23 (18.89) | 87.89 (11.62)

5. Secondary Outcome: Problem Areas in Diabetes Score
Description: Participants in the study report on daily problems with diabetes via this measure. Respondents indicate the degree to which each of the items is currently a problem for them. Score range: 0 to 4, higher scores correspond to more serious problems.
Time Frame: Baseline, 24 months
Population: Participants with complete data (by youth and parent) are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 49 | 21
score on a scale
  Youth - baseline: number analyzed (Participants) | 17 | 7
  Youth - baseline | 1.02 (0.72) | 0.78 (0.48)
  Youth - 24 months: number analyzed (Participants) | 17 | 7
  Youth - 24 months | 0.77 (0.81) | 0.43 (0.44)
  Parent - baseline: number analyzed (Participants) | 32 | 14
  Parent - baseline | 1.84 (0.73) | 2.11 (0.75)
  Parent - 24 months: number analyzed (Participants) | 32 | 14
  Parent - 24 months | 1.68 (0.75) | 1.74 (0.79)

6. Secondary Outcome: Diabetes Distress Scale
Description: This measure is widely used to capture the psychological distress experienced in relation to diabetes. Parent scale score range: 0-4. Youth scale score range: 1-6. Higher scores indicate greater diabetes-related distress.
Time Frame: Baseline, 24 months
Population: Participants with complete data (by youth and parent) are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 49 | 21
score on a scale
  Youth - baseline: number analyzed (Participants) | 17 | 7
  Youth - baseline | 1.87 (0.65) | 1.85 (0.67)
  Youth - 24 months: number analyzed (Participants) | 17 | 7
  Youth - 24 months | 1.85 (0.83) | 1.52 (0.46)
  Parent - baseline: number analyzed (Participants) | 32 | 14
  Parent - baseline | 1.19 (0.7) | 1.3 (0.6)
  Parent - 24 months: number analyzed (Participants) | 32 | 14
  Parent - 24 months | 1.32 (0.96) | 1.32 (1.05)

7. Secondary Outcome: Patient Health Questionnaire 9
Description: This is a widely used measure that captures depressive symptoms, and was used to assess health symptoms in parents. Score range: 0-24. Higher scores indicate greater severity of symptoms.
Time Frame: Baseline, 24 months
Population: Parent participants with complete data are included in the analysis. Youth did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 32 | 14
score on a scale
  Parent - baseline | 6.22 (5.52) | 9.22 (7.41)
  Parent - month 24 | 4.53 (4.53) | 3.71 (5.06)

8. Secondary Outcome: State-Trait Anxiety Inventory
Description: This is a widely used measure of anxiety symptoms, and was used to assess anxiety symptoms in parents. Score range for both state-anxiety is: 20-80. Higher scores indicate greater anxiety.
Time Frame: Baseline, 24 months
Population: Parent participants with complete data are included in the analysis. Youth did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 32 | 14
score on a scale
  Parent - baseline state-anxiety | 44.34 (11.84) | 49.71 (17)
  Parent - 24 months state-anxiety | 39.39 (14.87) | 34.05 (11.56)

9. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: This questionnaire measures the degree to which sleep is disrupted and the quality of sleep experienced by participants, and was used to assess sleep quality in parents. Score range is: 0-21. Higher scores indicate lower sleep quality.
Time Frame: Baseline, 24 months
Population: Parent participants with complete data are included in the analysis. Youth did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 32 | 14
score on a scale
  Parent - baseline | 7.04 (3.03) | 7.57 (3.9)
  Parent - 24 months | 6.1 (3.06) | 5.56 (2.96)

10. Secondary Outcome: Hypoglycemic Fear Survey
Description: People with diabetes worry about hypoglycemia, and was used to assess parent's worry about their child. This measure captures those worries. Score range: 0-72. Higher scores indicate greater fear and worry of hypoglycemia.
Time Frame: Baseline, 24 months
Population: Parent participants with complete data are included in the analysis. Youth did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 32 | 14
score on a scale
  Parent - baseline | 23.67 (12.56) | 23.86 (16.04)
  Parent - 24 months | 21.45 (15.42) | 19.62 (14.5)

11. Secondary Outcome: Hypoglycemic Confidence Questionnaire
Description: Hypoglycemia needs to be managed in various daily situations. This questionnaire captures confidence of the participants in those various situations, and was used to assess parent's confidence. Score range: 8-32. Higher scores indicate greater confidence to manage hypoglycemia.
Time Frame: Baseline, 24 months
Population: Participants with complete data (by youth and parent) are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 49 | 21
score on a scale
  Youth - baseline: number analyzed (Participants) | 17 | 7
  Youth - baseline | 23.65 (4.93) | 21.18 (5.55)
  Youth - 24 months: number analyzed (Participants) | 17 | 7
  Youth - 24 months | 26.92 (4.43) | 27.67 (8.81)
  Parent - baseline: number analyzed (Participants) | 32 | 14
  Parent - baseline | 19.46 (5.93) | 16.11 (6.21)
  Parent - 24 months: number analyzed (Participants) | 32 | 14
  Parent - 24 months | 24.9 (4.32) | 23.25 (5.31)

12. Secondary Outcome: General and Diabetes-specific Technology Use
Description: This measure has questions on attitudes and use of various general technologies (e.g., smartphone) and diabetes devices. Score range: 5-25. Higher scores indicate more positive attitudes about technology.
Time Frame: Baseline, 24 months
Population: Participants with complete data (by youth and parent) are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 49 | 21
score on a scale
  Youth - baseline: number analyzed (Participants) | 17 | 7
  Youth - baseline | 21 (2.4) | 19.71 (4.03)
  Youth - 24 months: number analyzed (Participants) | 17 | 7
  Youth - 24 months | 21.59 (2.7) | 21 (5.66)
  Parent - baseline: number analyzed (Participants) | 32 | 14
  Parent - baseline | 21.19 (3.04) | 20 (3.19)
  Parent - 24 months: number analyzed (Participants) | 32 | 14
  Parent - 24 months | 21.19 (3.8) | 21.92 (2.87)

13. Secondary Outcome: Center for Epidemiologic Studies Depression Measure
Description: This is a widely used measure of depression, and was used to assess depression symptoms in youths. Score range: 0-60. Higher scores indicate greater symptoms.
Time Frame: Baseline, 24 months
Population: Youth participants with complete data are included in the analysis. Parents did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 14 | 7
score on a scale
  Youth - baseline | 15.35 (10.28) | 9.57 (5.91)
  Youth - 24 months | 13.76 (12.44) | 10.64 (7.44)

14. Secondary Outcome: Child Health Utility 9D
Description: Widely used measure of quality of life that is used to generate quality-adjusted life years, and was used to assess health symptoms in youth. Each score scale is 0 to 4, with scores of 3 or 4 denoting more severe problems. The count of participants responding 3 or higher for each parameter are presented.
Time Frame: Baseline, 24 months
Population: Youth participants with complete data are included in the analysis. Parents did not complete this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 17 | 7
Participants
  Youth - baseline worried | 2 | 1
  Youth - 24 months worried | 0 | 0
  Youth - baseline sad | 2 | 1
  Youth - 24 months sad | 1 | 0
  Youth - baseline pain | 0 | 0
  Youth - 24 months pain | 1 | 0
  Youth - baseline tired | 4 | 0
  Youth - 24 months tired | 3 | 0
  Youth - baseline annoyed | 2 | 0
  Youth - 24 months annoyed | 1 | 0
  Youth - baseline schoolwork | 2 | 0
  Youth - 24 months schoolwork | 1 | 0
  Youth - baseline sleep | 1 | 1
  Youth - 24 months sleep | 0 | 0
  Youth - baseline routine | 0 | 0
  Youth - 24 months routine | 0 | 0
  Youth - baseline activities | 1 | 0
  Youth - 24 months activities | 1 | 0

15. Secondary Outcome: Hemoglobin A1c
Description: The hemoglobin A1c value is a biologic measure of the glycemia that is the gold standard measure of "control" of diabetes. Collected through a blood sample.
Time Frame: Baseline, 24 months
Population: Youth participants with complete data are included in the analysis. Parents are not included in this measure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 38 | 13
mg/dL
  Youth - baseline | 10.61 (2.02) | 10.64 (2.5)
  Youth - 24 months | 8.17 (1.77) | 7.5 (1.54)

16. Secondary Outcome: C-peptide
Description: This is a biologic measure of endogenous production and is collected through a blood sample.
Time Frame: Baseline, 24 months
Population: Youth participants with complete data are included in the analysis. Parent data was not collected.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CGM at Diagnosis of T1D | Usual Care
Number analyzed (Participants) | 31 | 12
ng/mL
  Youth - baseline | 0.66 (0.43) | 0.55 (0.29)
  Youth - 24 months | 0.14 (0.22) | 0.15 (0.17)

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events were assessed in youths only.
Arm/Group | CGM at Diagnosis of T1D | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/18
Other Adverse Events (participants affected / at risk) | 0/42 | 0/18

LIMITATIONS AND CAVEATS:
Primary and secondary survey outcome data is limited to participants with complete records.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT02734667/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT02734667/ICF_001.pdf